CLINICAL TRIAL: NCT04354597
Title: A Multicenter, Open-label, Pilot Study on Using Hydroxychloroquine (HCQ) and Azithromycin (AZ) Prophylaxis for Healthcare Workers With a Potential Risk of Exposure to COVID-19 Patients
Brief Title: Hydroxychloroquine and Azithromycin as Prophylaxis for Healthcare Workers Dealing With COVID19 Patients
Acronym: MOPHYDA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: New data not in favor of prophylaxis using this regimen
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Iyad Sultan, Chairman- Department of Pediatrics, Pediatrics Administration, King Hussein Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20 KHCC 67
Record Dates: First submitted 2020-04-09; First posted 2020-04-21 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; Prophylaxis; Hydroxychloroquine; Azithromycin
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Subjects who are enrolled in the study will be randomly assigned to any of the study arms, A or B.
  Study Arm A (HCQ & AZ)
  Study Arm B (No treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Arm A (HCQ & AZ) (Experimental): Subjects will receive weekly HCQ 400mg X 1 Day PO and AZ 500mg PO X 3 Days; weekly for 16 weeks.
  Interventions: Drug: HCQ & AZ
- Study Arm B (No treatment) (No Intervention): Subjects will receive no treatment in this group and will be serving as control.

INTERVENTIONS:
Drug: HCQ & AZ — Subjects will receive weekly HCQ 400mg PO and AZ PO 500mg X 3 Days; weekly for 16 weeks.
  Arms: Study Arm A (HCQ & AZ)

SUMMARY:
The main objective of this study is to assess the efficacy of the combination hydroxychloroquine and Azithromycin (HCQ and AZ) in reducing the infection risk among health care professionals in direct contact with COVID-19 patients.

DETAILED DESCRIPTION:
Exceptional efforts have been paid globally to apply the latest and most effective means of universal standard precautions throughout the settings facing COVID-19 crisis, and this is led by health care providers who are more vulnerable and have a higher risk of getting the infection (8.3% in Italy) and a higher rate of complications and mortality with some reports suggesting high mortality among these individuals.

While several clinical trials are underway across the globe to examine the effect of chloroquine at the moment, the number of COVID-19 cases is still on the rise and health care workers are facing a very high risk of getting the infection. In this study, we aim to study prophylactic efficacy of the combination (HCQ and AZ) among health care professionals in a 16 weeks period.

ELIGIBILITY:
Inclusion Criteria:

* Medical doctors, Nurses and Respiratory therapists caring for COVID-19 patients in ER and ICU and dedicated COVID19 units.
* Age between 18 and 70 years old.
* Male or non-pregnant, non- lactating female.
* Availability for follow up by phone.
* Willing to participate and provide signed informed consent.

Exclusion Criteria:

* Subjects with a history of retinopathy, sickle cell disease or trait, psoriasis, or porphyria.
* Subjects who take certain prescribed or over the counter (OTC) concomitant medication including ampicillin, cimetidine, digoxin, statins, cyclosporine, warfarin, fluconazole, within 2 weeks of dosing start, and during the duration of the study.
* Current Symptoms of Fever, Cough, or Shortness of Breath.
* PCR confirmed positive test of COVID-19.
* Weight < 40 kg.
* Pregnant (positive β-human chorionic gonadotropin test, β-HCG) or lactating female at the screening.
* Allergy to any of the study medications.
* History of splenectomy.
* Infection with hepatitis B or C viruses.
* Chronic or active neurologic disease including seizure disorder and chronic migraine headaches.
* Any abnormal baseline laboratory screening tests listed below

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)above twice the upper limit of normal for the reference lab.
  * Creatinine above the normal range.
  * Hemoglobin for males <12.5 g/dl and females <10.5 g/dl.
  * Platelet count of <150 X 103/L.
  * Total white blood cell (WBC) count out of normal range Note: If screening lab values are out of the normal range but are expected to be temporary (e.g. due to dehydration), they may be re-assessed one more time at the discretion of the investigator.
* An abnormal baseline screening ECG suggestive of cardiac disease as determined by a clinical investigator. QTcF of >450 msec for males and >470 msec for females.
* Any other significant finding that based on the judgment of the PI would increase the risk of having an adverse outcome from participating in this study
* Subjects known to have a mental illness
* Subjects who have Skin disorders (including rash, dermatitis, and psoriasis)
* Hematological disease.
* Cardiovascular disease.
* G6PD deficiency.
* Lactose intolerance.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Effect of HCQ and AZ in preventing infection with COVID-19 among healthcare workers working with COVID-19 patients | 4 Months
  Compare the proportion of participants who have RT-PCR confirmed infection with SARS-CoV-2 in both arms during the study period, measured by negative PCR test for SARS COV-2 virus

SECONDARY OUTCOMES:
Safety of HCQ and AZ | 4 Months
  Solicited and unsolicited adverse events in participants receiving HCQ+AZ during the study period, measured by the incidence of AEs in both arms. (The difference in type, number, and intensity)
Oxygen requirement | 4 Months
  The proportion of participants who require oxygen therapy for any indication during the study period in both arms, measured by the requirement for O2 or not in both arms.
ICU admission | 4 Months
  The proportion of participants who need ICU admission for any reason during the study period in both arms, measured by the incidence of ICU admission in both arms.
Mortality rate | 4 Months
  The proportion of participants who die of any cause during the study period in both arms, measured by the incidence of death in both arms.

CONTACTS AND LOCATIONS:
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided